CLINICAL TRIAL: NCT00579488
Title: Clinical Significance of Germline BRCA Mutations
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Cold Spring Harbor Laboratory (Other)
Responsible Party: Sponsor
Other Study IDs: 96-051
Record Dates: First submitted 2007-12-19; First posted 2007-12-24 (Estimated); Last update posted 2025-08-03 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer; Ovarian Cancer
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, Saliva, Buccal cell, Urine or Stool Tissue analysis and correlation of germline findings with somatic alterations within the tumor will be performed on a subset of individuals who have tumor tissue stored under protocol #06-107. Patients will be asked to fill out a baseline questionnaire on other medical, hormonal, and environmental risk factors.

SUMMARY:
The goal of this study is to help us learn more about the roles of genes in cancers that run in families. Sometimes, we are born with genes that are changed or altered. Gene changes are called mutations. Mutations may be passed down from parent to child. Some mutations cause a high risk for cancer. There are two major genes for breast and ovarian cancer. These genes are called BRCA --for breast cancer. If you have a mutation in these genes special actions may be needed. For a person with a known mutation, we will suggest ways to screen for cancer or prevent it. Not everything is known about cancer genes and mutations. The cancer screening we suggest may not always be effective. The aim of this study is to explore these questions. If you agree we will stay in touch with you to follow your medical history. We will also ask you about your family.

This will allow us to measure the cancer risks of known mutations. The study will also look for other cancer genes we do not know about. Whether or not you take part in this study, you may have gene testing. If you take part in this study and wish to know, we will tell your BRCA gene test results.

Beginning in 2019, a subset of participants will be given a follow-up questionnaire regarding their health and well-being.

The investigators may perform genetic testing on the blood or saliva sample in one of two ways: analysis for mutations in the BRCA1 and BRCA2 genes alone or as part of a panel of genes associated with breast cancer predisposition. New technologies are being employed for identification of patients with a susceptibility for developing breast cancer and thus analysis of multiple genes at one time may be offered to you. If this multi-gene testing applies to the patient, a question and answer sheet about this testing will be provided to them by their genetic counselor.

ELIGIBILITY:
Inclusion Criteria:

* Families referred for genetic counseling consultation at Memorial Hospital
* Individuals self-referred or physician referred for genetic counseling due to a concern about increased risk for breast cancer, regardless of family history or ethnic origin.
* Individuals enrolled in MSK protocol 97-029 "Germline BRCA1 and BRCA2 mutations in Jewish Women Affected by Breast Cancer"
* Individuals who present for genetic counseling consultation at Memorial Hospital after undergoing genetic testing at an outside institution.
* Member of a family with breast cancer who wishes to provide a DNA sample for research purposes
* Individuals enrolled on protocol 12-245 with germline variants in genes associated with risk for breast or ovarian cancer, or absent such variants in the presence of a family history or other phenotypic features of interest including but not limited to: triple negative breast cancer, early onset of disease, and/or synchronous or metachronous breast and ovarian cancer.

Exclusion Criteria:

-Patients will be excluded from this study if: he/she has physical, cognitive or psychiatric conditions that interfere with ability to give meaningful informed consent; he/she cannot read, write or communicate in English; he/she is less than 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary Care Clinic
Sampling Method: Non-Probability Sample
Enrollment: 13320 (Actual)
Dates: Start 1996-07; Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
To obtain DNA samples | 2 years
  for the purpose of estimating relative risk of BRCA1 ,BRCA2 and other gene mutations for breast cancer incidence in families with breast or ovarian cancer.

SECONDARY OUTCOMES:
To obtain clinical and follow-up information on individuals being tested for BRCA mutations, in order to assess penetrance & phenotypic correlations of specific mutations, & to describe the outcome of medical or surgical interventions in heterozygotes. | 2 years
To establish a confidential registry/repository containing data on specific mutations and genomic variants and clinical feature as well as DNA for future gene discovery. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Offit, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

REFERENCES:
- See also: Related Info — http://www.mskcc.org